CLINICAL TRIAL: NCT04484545
Title: Prognostic Factors in Patients Admitted to an Urban Teaching Hospital With COVID-19 Infection
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Glasgow Royal Infirmary (Other)
Responsible Party: Principal Investigator, Dr. Donogh Maguire, Emergency Medicine Consultant, Glasgow Royal Infirmary
Other Study IDs: IRAS 282807
Record Dates: First submitted 2020-07-22; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alive or Dead with COVID-19 diagnosis: Patients selected in phase 1 of study according to Health Protection Scotland criteria for diagnosis of COVID-19 infection Patients selected for phase 2 (validation phase) by PCR result
  Interventions: Diagnostic Test: Prognostic score

INTERVENTIONS:
Diagnostic Test: Prognostic score — Validation of scores of systemic inflammatory response

SUMMARY:
As of 27th May 2020, approximately 5.7 million people worldwide are known to have been infected with COVID-19 coronavirus and more than 350,000 have died (1). The severity of this viral disease for an individual is associated with a widespread perturbation of immune, physiological and metabolic parameters (2, 3). These whole body changes could be considered characteristic of a systemic inflammatory response to tissue injury and it has been long recognised that a large and ongoing systemic inflammatory response is associated with the development of multiple organ failure and infective disease (4, 5).

One of the cardinal signs of severe COVID-19 infection is a marked systemic inflammatory response (2). This response bears striking similarity to the systemic inflammatory response experienced by patients undergoing major elective surgical resections for cancer (6, 7). Indeed, the systemic inflammatory response and the associated metabolic stress has been most well characterised in major elective surgery, where the relationship between the magnitude of the post-operative systemic inflammatory response and the development of post-operative complications is now well recognised, as is the effect of patient comorbidity on this relationship (8, 9). Such work has informed therapeutic manoeuvres including minimally invasive surgery, pre-operative optimisation (e.g. anaesthesia, nutrition and steroids) and enhanced recovery protocols.

The aim of the present study was to examine whether routinely collected clinicopathological characteristics of patients with COVID-19 on admission were informative on the immune and metabolic stress experienced by patients with COVID-19 and whether such characteristics were informative on subsequent outcome.

DETAILED DESCRIPTION:
Electronic patient records for patients who attended the Emergency Department (ED) and Acute Assessment Unit (AAU) at Glasgow Royal Infirmary (GRI), Glasgow, U.K., during the initial 7-week period of the COVID-19 pandemic in Glasgow city (17th March 2020 - 1st May 2020) were examined for routine clinical, laboratory and clinical outcome data. GRI is a university teaching hospital that serves an urban population with a high burden of socio-economic deprivation and offers the full spectrum of adult acute receiving specialties to patients over 16 years old. In line with NHS policy, this study was approved by the NHS Greater Glasgow and Clyde Caldicott guardian.

ELIGIBILITY:
Inclusion Criteria:

* Clinical, radiological and PCR positive COVID-19 diagnosis

Exclusion Criteria:

* less than 18 years old

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General hospital population
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
mortality | 30-day
  30-day mortality and prognostic score

CONTACTS AND LOCATIONS:
Overall Officials: Donogh Maguire, PhD, Principal Investigator — NHS GGC
Locations (1):
- Glasgow Royal Infirmary, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised patient data will be made available on reasonable request
Supporting Information: CSR
Time Frame: 6 months

REFERENCES:
- [Derived] McGovern J, Al-Azzawi Y, Kemp O, Moffitt P, Richards C, Dolan RD, Laird BJ, McMillan DC, Maguire D. The relationship between frailty, nutritional status, co-morbidity, CT-body composition and systemic inflammation in patients with COVID-19. J Transl Med. 2022 Feb 21;20(1):98. doi: 10.1186/s12967-022-03300-2. PMID 35189900
- [Derived] Maguire D, Richards C, Woods M, Dolan R, Wilson Veitch J, Sim WMJ, Kemmett OEH, Milton DC, Randall SLW, Bui LD, Goldmann N, Brown A, Gillen E, Cameron A, Laird B, Talwar D, Godber IM, Wadsworth J, Catchpole A, Davidson A, McMillan DC. The systemic inflammatory response and clinicopathological characteristics in patients admitted to hospital with COVID-19 infection: Comparison of 2 consecutive cohorts. PLoS One. 2021 May 27;16(5):e0251924. doi: 10.1371/journal.pone.0251924. eCollection 2021. PMID 34043668